CLINICAL TRIAL: NCT00001027
Title: A Phase I/II Trial of Parenteral Pentamidine for PCP Prophylaxis in HIV-Infected Children Who Are Intolerant to Oral Trimethoprim-Sulfamethoxazole
Brief Title: A Study of Pentamidine in the Prevention of Pneumocystis Carinii Pneumonia (PCP) in HIV-Infected Children Who Cannot Take Trimethoprim-Sulfamethoxazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Fujisawa Pharmaceutical Co (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 189; 11164 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Pneumonia, Pneumocystis carinii; Pentamidine; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Pentamidine

INTERVENTIONS:
Drug: Pentamidine isethionate

SUMMARY:
Primary: To compare the pharmacokinetics of biweekly and monthly dose regimens of intravenous pentamidine in HIV-infected infants and children who require PCP prophylaxis and who are intolerant to oral trimethoprim - sulfamethoxazole. To determine the safety and tolerance of these regimens in this patient population.

Secondary: To obtain information on the rate of PCP breakthrough in infants and children receiving parenteral pentamidine prophylaxis.

Prophylaxis against Pneumocystis carinii pneumonia is recommended for all HIV-infected children considered to be at high risk. In children younger than 5 years of age with intolerance to trimethoprim - sulfamethoxazole, parenteral pentamidine may be a successful alternative.

DETAILED DESCRIPTION:
Prophylaxis against Pneumocystis carinii pneumonia is recommended for all HIV-infected children considered to be at high risk. In children younger than 5 years of age with intolerance to trimethoprim - sulfamethoxazole, parenteral pentamidine may be a successful alternative.

Thirty-two children are randomized to one of two treatment arms. Patients receive pentamidine on either a biweekly or a monthly treatment schedule. Treatment continues until the last child enrolled has received at least 6 months of pentamidine. Patients are stratified according to age < 24 months or age >= 24 months. Steady-state pharmacokinetics will be examined in a subsample of 20 patients.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Steroids and intravenous immune globulin (IVIG).

Patients must have:

* Documented HIV infection.
* Need for PCP prophylaxis.
* Known intolerance to trimethoprim - sulfamethoxazole (TMP-SMX).

One of the following required conditions:

* Known intolerance or allergy to dapsone; G6PD deficiency; history of serious or life-threatening reaction to TMP-SMX; exclusion from protocol ACTG 179; election by parent not to enroll child on ACTG 179; or receiving medical care at sites not participating in ACTG 179.

NOTE:

* Co-enrollment in other ACTG pediatric studies is permitted.

Consent of parent or guardian is required.

Prior Medication:

Allowed:

* Prior pentamidine.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Active PCP.
* Pancreatitis defined as amylase elevation associated with an elevated lipase that is > 2 x upper limit of normal.

Prior Medication:

Excluded:

* TMP-SMX or dapsone within 7 days prior to study entry (toxicities to TMP-SMX or dapsone must be clearly resolving).

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32
Dates: Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Van Dyke R, Study Chair; Pramberg J, Study Chair
Locations (13):
- United States (11):
  - Usc La Nichd Crs, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - SUNY Upstate Med. Univ., Dept. of Peds, Syracuse, New York
- Puerto Rico (2):
  - San Juan City Hosp. PR NICHD CRS, San Juan
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan